CLINICAL TRIAL: NCT05751486
Title: A Randomised, Open-label, Phase I Dose Exploration Study to Compare Single, Multiple, and Long-term Dosing of Toripalimab Injection (Subcutaneous) With Toripalimab Injection (IV) in Patients With Advanced Nasopharyngeal Carcinoma
Brief Title: A Clinical Study to Evaluate the Safety and Tolerability of JS001sc in Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS001sc-001-I
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JS001sc Q3W (Experimental)
  Interventions: Biological: Toripalimab injection(subcutaneous)/JS001sc
- JS001sc long period (Experimental)
  Interventions: Biological: Toripalimab injection(subcutaneous)/JS001sc
- JS001 IV (if applicable) (Experimental): the Safety Monitor Committe (SMC) will discuss whether to conduct an IV cohort and determine the dose/frequency of the IV cohort, based on the initial safety and clinical pharmacological data of triprilimab injection in combination with the GP regimen;
  Interventions: Biological: Toripalimab /JS001
- Additional cohort (if applicable) (Experimental): The exploration of additional dosing/frequency will be discussed by the SMC based on prior safety and clinical pharmacological data
  Interventions: Biological: Toripalimab injection(subcutaneous)/JS001sc

INTERVENTIONS:
Biological: Toripalimab injection(subcutaneous)/JS001sc — JS001sc Q3W combination with gemcitabine and cisplatin.
  Arms: JS001sc Q3W
Biological: Toripalimab injection(subcutaneous)/JS001sc — JS001sc long period combination with gemcitabine and cisplatin.
  Arms: JS001sc long period
Biological: Toripalimab /JS001 — JS001 IV (if applicable) .
  Arms: JS001 IV (if applicable)
Biological: Toripalimab injection(subcutaneous)/JS001sc — Additional cohort (if applicable)
  Arms: Additional cohort (if applicable)

SUMMARY:
The purpose of this phase I clinical study was to evaluate the safety and tolerability of JS001sc monotherapy and combination with gemcitabine and cisplatin (GP) in patients with Advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This study is the first human study of Toripalimab injection(subcutaneous) .Patients with advanced nasopharyngeal carcinoma were planned to be enrolled.

Two cohorts were initially proposed, Toripalimab injection (subcutaneous) Q3W combination with gemcitabine and cisplatin (GP) regimen and JS001sc long-term dosing combined with GP regimen.

Cohort 1: JS001sc Q3W SC combined with GP regimen chemotherapy; Cohort 2: JS001sc long period SC combined with GP regimen chemotherapy; IV cohort (if applicable): the Safety Monitor Committe (SMC) will discuss whether to conduct an IV cohort and determine the dose/frequency of the IV cohort, based on the initial safety and clinical pharmacological data of triprilimab injection in combination with the GP regimen; Additional cohort (if applicable): the exploration of additional dosing/frequency will be discussed by the SMC based on prior safety and clinical pharmacological data.

Subjects with no disease progression (PD) after the combination chemotherapy period (JS001/JS001SC combined with GP regimen, in one therapeutic cycle of three weeks, for at most 6 cycles) will enter the monotherapy maintenance period.JS001/JS001sc monotherapy maintenance treatment of the same dose/frequency f the combination chemotherapy period.Based on the preliminary safety and clinical pharmacological data, SMC will discusses whether to change the dose/frequency.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study with full informed consent and signed written informed consent form;
2. Recurrent/metastatic nasopharyngeal carcinoma diagnosed histologically and/or cytologically,Patients with no loco-regional therapy or radical therapy of primary metastatic （UICC&AJCC 8th edition) or recurrent nasopharyngeal carcinoma after radical therapy.No previous systematic treatment for recurrent or metastatic disease.
3. Patients with recurrent nasopharyngeal carcinoma after radical therapy must be satisfied that the disease recurrence more than 6 months after the last radiotherapy or chemotherapy.
4. There should be at least one measurable lesion according to RECIST V1.1 evaluation criteria. The lesions that have previously received radiotherapy should not be considered as target lesions unless there is definite progression after radiotherapy.
5. Age of 18-75 years (inclusive), male or female;
6. The physical status score is 0 or 1 on the Eastern Oncology Collaboration (ECOG) scale;
7. The expected survival is ≥3 months;
8. Major organ functions meet the following requirements.No blood transfusion or blood products, hematopoietic stimulating factors or other drugs were used to correct blood cell counts within 14 days prior to the examination：

   Neutrophil absolute count ≥1.5 × 109/L;

   Platelet count ≥ 100 × 109/L;

   Hemoglobin ≥ 90 g/L;

   Serum albumin ≥ 30 g/L;

   Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) with biliary obstruction resolved prior to randomization;

   Alkaline phosphatase (ALP)≤ 3 × ULN, ALP≤ 5 × ULN (Patients may have liver or bone metastasis);

   Albumin ≥ 30 g/L;

   Serum creatinine (Cr) ≤ 1.5 × ULN, Cr clearance ≥ 60 mL/min (Cockcroft -Gault Formulas, refer to attachment 2);

   International Normalized Ratio (INR), prothrombin time (PT), and activated Partial thrombin Time (aPTT) ≤ 1.5× ULN (Patients should not have received anticoagulant therapy);If Patients receiving anticoagulant therapy that they should use a steady dose;
9. Within 7 days prior to the first dose, women of reproductive age must be confirmed as having a negative serum pregnancy test and consent to use effective contraception during the duration of study drug use and for 150 days after the last dose. Women of childbearing age are defined as sexually mature women: 1) no hysterectomy or bilateral ovariectomy, 2) Natural menopause did not last for 24 consecutive months (Amenorrhea after cancer treatment does not rule out fertility);Male patients with a female partner of reproductive age agreed to use effective contraception during the study drug use period and for 6 months after the last dose;

Exclusion Criteria:

1. A history of severe allergic reactions to to any component of JS001;
2. A history of hypersensitivity to gemcitabine or cisplatin or any excipients;
3. Prior treatment with Anti-PD-1 antibody, anti-PD-L1 or anti-CTLA-4 antibody;
4. Received antitumor therapy ,Such as, chemotherapy, radiotherapy,immune therapy therapy, biological drugs therapy or other investigational drugs within 4 weeks or 5 half-lives period （Choose the shorter one）before the administration of the first dose;Receive traditional Chinese medicine or Chinese patent medicine preparations with anti-tumor indications within 2 weeks prior to initial administration;
5. Within 28 days prior to the first study drug administration, there are other major surgeries except for the diagnosis of nasopharynx carcinoma, or assessed by researchers and specialists that they did not have fully recovered from the complications of major surgery;
6. The toxic response of previous anti-tumor treatment has not been restored to CTCAE 0-1, except for hair loss and pigmentation.Irreversible toxicity reasonably expected not to be aggravated by the drug under study (e.g. hearing loss). They can be included after confirmation with the sponsor.
7. A subject with clinical symptoms of CNS and/or cancer meningitis (such as cerebral edema, hormone intervention, or brain metastases) No clear surgery and/or radiotherapy for spinal cord compression, or for spinal cord compression that previously diagnosed and treated, no evidence indicates that the first study of pre -dating diseases in clinical stability ≥2 weeks of clinical clinic; Received the treatment of brain or meningeral membrane, such as clinical stability has been maintained for at least 2 months, and has stopped systemic hormone therapy (dose> 10 mg/day dawnone or other curative hormones such as);
8. Poorly controlled the thoracic effusion, pericardial effusion, or ascites that need to be drained (thoracic ascites ≥1 times/month)
9. Poorly controlled tumor-related pain:

   For patients who need analgesic treatment, they must receive a stable dose treatment before participating in the study ; Before entering the group, a clinical indication lesions should be treated for local treatment (for example, bone metastases or metastasis of neurotransidal);
10. Featured pulmonary fibrosis, drug -induced pneumonia, mechanized pneumonia (that is, occlusion fine pineitis), radioactive pneumonia with clinical symptoms or steroids, active pneumonia or other medium -weight lungs that seriously affect lung function that seriously affect lung function disease;
11. The first 4 weeks before the medication found that there were necrotic lesions, and the researchers judged that there was a risk of hemorrhage;
12. Within the first 5 years of administration, there are other malignant tumors other than nasopharyngeal cancer (except for cured cervical in situ cancer, base or squamous cell skin cancer, limited prostate cancer or Ductal carcinoma in situ of breast);
13. The subject has any active autoimmune disease or a history of autoimmune diseases within two years. Except for the following situations: 1) patients with thyroid dysfunction, receiving stable dose thyroid hormone replacement treatment; 2) receiving stable insulin therapy schemes Later, patients with type I diabetes were obtained; 3) skin diseases that do not need to be treated with whole body, such as psoriasis, vitiligo, etc. (for more comprehensive list of autoimmune diseases, see Annex 4);
14. Severe infections (CTCAE> 2) within 28 days before the administration (CTCAE> 2), such as severe pneumonia, fungal ledis, infection complications, etc. that need to be hospitalized;
15. Availability with active lung tuberculosis (TB) is undergoing anti -tuberculosis treatment or screening within one year before receiving anti -tuberculosis treatment;
16. It suffers from corticosteroids that require long -term use of immunosuppressive drug treatment, or the use of immunosuppressive dose (dose> 10 mg/day or other curative hormones such as 10 mg/day);
17. Received any live vaccine within 4 weeks before the medication (for example, vaccines for infectious diseases, such as influenza vaccines, chickenpox vaccines, etc.);
18. Women of pregnancy or lactation;
19. Known human immune defect virus (HIV) positive patients;
20. Hepatitis B core antibodies (HBCAB) or hepatitis B surface antigen (HBSAG) positive detection of HBV DNA copy number ≥1000CPS/ml or reference value limit;
21. Hepatitis C (HCV) antibody positive at the same time detected HCV RNA copies of positive;
22. Patients who have been transplanted in the same kind of album bone marrow or previously performed physical organ transplantation;
23. There are severe nerve or mental illness, including dementia and seizures;
24. Due to NCI-CTCAE ≥ 2 peripheral neuropathy;
25. With major cardiovascular diseases, such as the New York Heart Diseases (NYHA) heart function grading II or above heart disease (see Annex 3), the myocardial infarction and control within 3 months before the first study; Unstable angina pectoris; Knitrines of patients with coronary arteries, congestive heart failure of the above standards, or left ventricular ejection scores <50%of patients must use the optimized stable medical plan determined by the doctor. If appropriate, you can consult the heart. Sick expert;
26. Investigators are judged that they are not suitable for other situations in this study, including but not limited to any disease or medical history that may confuse the results o study and interfere with patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | At designated time points (Approximately 2 years)
  Maximum observed serum concentration
Tmax | At designated time points (Approximately 2 years)
  Time of maximum observed serum concentration
AUC | At designated time points (Approximately 2 years)
  Area Under the Concentration-Time Curve
CL | At designated time points (Approximately 2 years)
  Clearance
Volume of Distribution | At designated time points (Approximately 2 years)
  V
F | At designated time points (Approximately 2 years)
  Bioavailability
Ctrough | At designated time points (Approximately 2 years)
  Trough observed serum toripalimab concentration

SECONDARY OUTCOMES:
Immunogenicity | Up to approximately 24 months from first patient in.
  Incidence of anti-drug antibody (ADA) and/or neutralizing antibody (Nab), titer of ADA positive samples
adverse events (AE), immune-related adverse events (irAE) and serious adverse events (SAE) | Until 2 years after the last subject was enrolled
  To evaluate incidence, severity and outcome of adverse events (AE), immune-related adverse events (irAE) and serious adverse events (SAE)
ORR | Up to approximately 24 months from first patient in.
  Objective response rate (ORR) was assessed based on RECIST V1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No